CLINICAL TRIAL: NCT06083350
Title: A Randomized Controlled Trial of Yeast Beta-glucan on Cognitive Function in Patients With Mild Cognitive Impairment
Brief Title: Effects of Yeast Beta-glucan on Cognitive Function in Patients With Mild Cognitive Impairment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaofan Xu (Other)
Responsible Party: Sponsor-Investigator, Xiaofan Xu, Principal Investigator, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HuazhongU-XXu
Record Dates: First submitted 2023-09-26; First posted 2023-10-16 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
Keywords: Mild Cognitive Impairment; Alzheimer Disease; Montreal Cognitive Assessment; Gut microbiota
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple blind, the unique codes of the intervention and placebo are known only to the person in charge of the intervention manufacturer (Anginute), not to the study implementors, investigators, subjects, data collectors and analysts, and are only unblinded by the manufacturer after the study is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yeast beta-glucan (Experimental): Yeast beta-glucan capsules, 250mg，taken with meals, two capsules twice a day
  Interventions: Dietary Supplement: Yeast beta-glucan
- Starch (Placebo Comparator): Starch capsule, 250mg, taken with meals, two capsules twice a day
  Interventions: Dietary Supplement: Starch

INTERVENTIONS:
Dietary Supplement: Yeast beta-glucan — Produced by Angel Yeast Co., LTD
  Arms: Yeast beta-glucan
Dietary Supplement: Starch — Produced by Angel Yeast Co., LTD
  Arms: Starch

SUMMARY:
Patients with mild cognitive impairment aged 50-80 years old were recruited in Shiyan City, Hubei Province, and divided into intervention group and placebo group. They were given yeast β-glucan capsules and starch capsules, respectively, for 6 months, in order to explore whether yeast β-glucan can improve cognitive function of patients with mild cognitive impairment by regulating gut microbiota and its metabolites.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 50-80 years;
* 2. Permanent residents of Shiyan City;
* 3. Meet the diagnostic criteria of MCI:
* 4. Willing to cooperate in completing questionnaire survey and clinical examination, and sign informed consent;
* 5. Did not participate in other clinical trials in the past 3 months.

Exclusion Criteria:

* 1. Alcohol or drug abuse;
* 2. Patients with neurological diseases that may cause cognitive dysfunction, including cerebrovascular diseases, stroke, brain tumors, Parkinson's disease, active epilepsy, etc.;
* 3. History of severe head trauma;
* 4. Severe sensory and perceptual impairment, unable to complete the cognitive function measurement;
* 5. History of mental illness such as depression, mania, anxiety, or take psychiatric drugs;
* 6. Serious heart, lung, liver, kidney dysfunction, malignant tumors, etc.;
* 7. Suffering from autoimmune diseases;
* 8. Trauma, spinal injury or any disease that may affect the motor function of the limb;
* 9. Recent infectious diseases, acute gastrointestinal diseases;
* 10. Take antibiotics, probiotics, prebiotics or biostime products within the last 1 month.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment, MOCA | up to 7 months
  To assess overall cognitive function based on test scores. Patients with MOCA scores between 18 and 25 were included, and higher scores mean a better outcome.

SECONDARY OUTCOMES:
Gut microbiota, fecal SCFAs and SIgA | up to 2 years
  16S rRNA gene amplicon sequencing technique is used to determine species richness and diversity, species difference and functional prediction of gut microbiota; The content of SCFAs in fecal is determined by gas chromatography-mass spectrometry (GC-MS); Fecal SIgA is detected by enzyme-linked immunosorbent assay (ELISA).
T/B/NK cells and IL-1β，IL-2，IL-4，IL-5，IL-6，IL-8，IL-10，IL-12p70，IL-17，IFN-γ and TNF-α in peripheral blood | up to 7 months
  The types and absolute counts of T/B/NK cells in peripheral blood are detected by flow cytometry, Plasma levels of IL-1β, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12p70, IL-17, IFN-γ, and TNF-α are measured by Cytometric Bead Array (CBA) technology.
Plasma Aβ-40, Aβ-42 | up to 2 years
  The plasma levels of Aβ-40 and Aβ-42 were detected by ELISA
Clock Drawing Test | up to 7 months
  To assess visual space and executive ability. Higher scores mean a better outcome.
Digital Span Test | up to 7 months
  Attention and short-term memory are assessed by Digital Span Test. Higher scores mean a better outcome.
Trail Making Test | up to 7 months
  To assess visual space and executive ability. The shorter the time, the lower the error rate, and the better the result.
Verbal Fluency Test | up to 7 months
  To assess verbal fluency. Higher scores mean a better outcome.
Digit Symbol Substitution Test | up to 7 months
  To assess reaction speed. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofan Xu, Master, Principal Investigator — School of Public Health, Tongji Medical College, Huazhong University of Science and Technology
Locations (2):
- China (2):
  - Sinopharm Dongfeng General Hospital, Shiyan, Hubei
  - Huazhong University of Science and Technology, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No